CLINICAL TRIAL: NCT01292668
Title: A Phase I Study for Superficial Basal Cell Carcinoma to Determine the Irradiance - Dependent Pain Threshold for Methylaminolevulinate (MAL)/PDT.
Brief Title: Photodynamic Therapy Using Methyl-5-Aminolevulinate Hydrochloride Cream in Determining Pain Threshold in Patients With Skin Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 175410; NCI-2010-02319 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Basal Cell Carcinoma of the Skin; Pain; Recurrent Skin Cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Pain; Skin Neoplasms | interventions — Photochemotherapy; 1-phenyl-3,3-dimethyltriazene; Laser Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (Experimental): Patients apply methyl-5-aminolevulinate hydrochloride (MAL) cream on the lesions and the surrounding normal skin. Beginning 3 hours later, patients undergo laser light treatment for 3-5 minutes.
  Interventions: Drug: methyl-5-aminolevulinate hydrochloride cream; Procedure: laser therapy
- Group II (Experimental): Patients apply MAL cream on the lesions and the surrounding normal skin. Beginning 3 hours later, patients undergo light emitting diode treatment for 5-10 minutes.
  Interventions: Drug: methyl-5-aminolevulinate hydrochloride cream; Drug: photodynamic therapy

INTERVENTIONS:
Drug: methyl-5-aminolevulinate hydrochloride cream — Applied topically
  Other Names: Metvix cream; Metvixia cream
Drug: photodynamic therapy — Undergo light-emitting diode photodynamic therapy
  Other Names: Light Infusion Therapy™; PDT; therapy, photodynamic
  Arms: Group II
Procedure: laser therapy — Undergo laser light photodynamic therapy
  Other Names: therapy, laser
  Arms: Group I

SUMMARY:
RATIONALE: Photodynamic therapy uses a drug that becomes active when it is exposed to a certain kind of light. When the drug is active, cancer cells are killed. Photodynamic therapy using methyl-5-aminolevulinate hydrochloride cream may be effective against skin cancer. PURPOSE: This phase I trial is studying the side effects and best dose of photodynamic therapy with methyl-5-aminolevulinate hydrochloride cream in determining pain threshold patients with skin cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES: I. To determine the "low" initial irradiance that causes no or minimal (pain grade of < 4) during the time period during which 90 +/- 10% photo bleaching of protoporphyrin IX (PplX) in the lesion occurs, and which precedes the "high" irradiance portion of MAL/PDT. II. To determine the effects of preceding "low" irradiance on the pain level of the "high" irradiance portion of MAL-PDT. SECONDARY OBJECTIVES: I. To determine the effects of irradiance on lesion perfusion. II. To determine PpIX and Total Vit D content in blood. TERTIARY OBJECTIVES: I. To monitor the clinical outcomes of the treatments for initial response and recurrences. OUTLINE: Patients are randomized to 1 of 2 treatment arms. GROUP I: Patients apply methyl-5-aminolevulinate hydrochloride (MAL) cream on the lesions and the surrounding normal skin. Beginning 3 hours later, patients undergo laser light treatment for 3-5 minutes. GROUP II: Patients apply MAL cream on the lesions and the surrounding normal skin. Beginning 3 hours later, patients undergo light-emitting diode treatment for 10-20 minutes. After completion of study treatment, patients are followed up at 5-7 days, at 6-12 months, and at 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 1-2 superficial basal cell carcinoma (sBCC), 0.5 to 2 cm in diameter
* Primary or recurrent lesions may be treated
* Diagnosis must be confirmed by biopsy, at least 2 weeks pre treatment
* Each patient with < 8 lesions can contribute a maximum of 2 lesions per treatment session, 1 lesion per light source, which can be treated the same day as permitted by scheduling; the remaining lesions may be treated as soon as scheduling permits with non protocol Photodynamic Therapy
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Patients not meeting the above selection criteria
* Lesions which are not suitable for diagnostic measurements
* Patients with >= 8 lesions to be treated
* Carcinomas of types known to have uncertain clinical margins (e.g. morpheaform or infiltrating), or any lesion felt to require Mohs surgery for definitive control
* Lesions over boney prominences
* Patients with porphyrias or known hypersensitivity to porphyrins
* Patients with known photosensitivity diseases
* Patients with allergies to Metvixia (MAL) cream ingredients (peanut and almond oil)
* Patients previously treated with a systemic photo sensitizer within 4 months
* Pregnant or nursing female patients
* Patients unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Irradiance-dependent pain threshold | 30-60 sec after the initial "low" irradiance treatment, every 3-5 min until irradiance increase, 30-60 sec after the "high" irradiance increase, and every 3-5 min until end of treatment

SECONDARY OUTCOMES:
Efficacy of treatment in terms of clinical response | At 5-7 days, at 6-12 months, and at 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Ilene L Rothman, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States